CLINICAL TRIAL: NCT05463718
Title: Virtual Reality Versus Balance Beam on Walking Performance in Children With Spastic Hemiplegic Cerebral Palsy
Brief Title: Virtual Reality Versus Balance Beam on Spastic Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohanad Mohsen Madboly Elsayed, Principal Investigator, Pediatrics department, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003683
Record Dates: First submitted 2022-06-19; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-01

CONDITIONS: Balance Problems in Spastic Hemiplegic Children; Walking Performance in Spastic Hemiplegic Children

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- children treated by the traditional physical therapy program based on Neurodevelopmental technique (Experimental): Twenty-five cerebral palsied hemiplegic children will be treated by the traditional physical therapy program ( balance board, single limb support, standing with throwing ball ) based on Neurodevelopmental technique for 6 month
  Interventions: Device: Virtual Reality
- children treated by Virtual Reality for 15 min. besides the traditional physical therapy program (Experimental): twenty-five cerebral palsied hemiplegics will be included in this group; they will be receive the regular physical therapy program in addition to training by Virtual reality with use of the HMD helmet allows users to perceive a 3D stereoscopic images that enable participants to interact with different balance games as football Soccer, football heading (known as Soccer Heading), the tight rope walks and the Penguin slide game.
  Interventions: Device: Virtual Reality
- children treated by Balance Beam for 15 min besides the traditional physical therapy program (Experimental): Twenty-five cerebral palsied hemiplegics will be included in this group; they will be receive the regular physical therapy program in addition to training by standing and walking in balance beam by differentiate levels of walking balance proficiency as varying widths of beam and walking in different direction (forward or backward).
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — children treated by Virtual Reality for 15 min. besides the traditional physical therapy program

SUMMARY:
Is there any difference between the use of Virtual reality and Balance beam on walking performance in children with Spastic Hemiplegic Children?

DETAILED DESCRIPTION:
To compare the effect of Virtual reality and the traditional physical therapy program based on Neurodevelopmental technique with Spastic Hemiplegic Children.

To compare the effect of Balance beam and the traditional physical therapy program based on Neurodevelopmental technique with Spastic Hemiplegic Children.

To compare the effect of Virtual reality and Balance beam on walking performance in children with Spastic Hemiplegic Children.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 7 to 11 years old, from both genders.
* Modified Ashworth scale adopted from, (Bohannon and Smith,1987) was used to select the patients with grade 1 and 1+ of Spasticity.
* They were able to stand and walk.
* Gross motor function measure scale GMFM (level I &II). (Russell et al. ,2013).
* Children with good mentality to understand the evaluation steps.

Exclusion Criteria:

* Children who have orthopedic surgery or Botulinum Toxin-A injection in the last 6 months.
* Children who have any spinal deformities.
* Children with severe muscle contracture.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Balance it will be assist by HUMAC Balance Assessment system | 6 month
  Evaluation materials that used in assist balance :
  HUMAC Balance Assessment system consists of:
  1- The force platform 2- The HUMAC CD holding the operating program This test will be use assess the sensory integration of balance and postural control in the conditions of eyes open and eyes closed from standing, lasts for 30 second and the test was repeated for three times and the mean value is calculated from the result of each trial which appears in the form of percent of stability in each trial
Walking ability | 6 month
  Evaluation materials
  Six Minute Walk Test (6MWT) it is a valid and reliable instrumentation using to asses walking capacity The child of this test is to walk as far as possible for 6 minutes. You will walk back and forth in this hallway, after the test, measured walking capacity exercise (BP, HR and SpO2) were re-measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Cairo, Egypt